CLINICAL TRIAL: NCT06536920
Title: Frequency and Impact of Migraine Among Sohag University Students
Brief Title: Migraine Among Sohag University Students
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Ahmed ElSayed Sadek, Principle investigator, Sohag University
Other Study IDs: Soh-24-05-03MS
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Sohag university students: Who diagnosed as migraine among sohag university students
  Interventions: Diagnostic Test: Migraine screening questionnaire

INTERVENTIONS:
Diagnostic Test: Migraine screening questionnaire — Screening test

SUMMARY:
Diagnosis of migraine among students and detect frequency among them and detect how far migraine affect their life

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 25 years old.
* students accept to give informed consent

Exclusion Criteria:

* Students refused to give informed consent
* Age less than 18 or more than 25 ears old.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Sohag university students
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Migraine screening questionnaire | 1 year
  Knowing frequency of migarine and impact of migraine on students' normal life

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt